CLINICAL TRIAL: NCT06369259
Title: Open-label Phase 2 Study of Avutometinib (RAF/MEK Clamp) in Combination With Defactinib (FAK Inhibitor) and Cetuximab in Patients With Unresectable, Anti-EGFR-Refractory Advanced Colorectal Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023-0997; NCI-2024-03302 (Other: NCI-CTRP Clinical Registry)
Record Dates: First submitted 2024-04-12; First posted 2024-04-16 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Advanced Colorectal Cancer
MeSH Terms: interventions — defactinib; Cetuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Safety Run In (Experimental): If you are enrolled in the Safety Run In group, the dose of avutometinib you receive will depend on when you join this study. Up to 3 dose levels of avutometinib will be tested, and between 3-6 participants will be enrolled at each dose level.
  The first group of participants will receive the planned starting dose level of avutometinib. Then, if no intolerable side effects are seen, a second group of participants will be enrolled to receive a higher dose. If intolerable side effects are seen, the second group will receive a lower dose. One of these 3 doses will be selected as the recommended dose of avutometinib in combination with cetuximab and defactinib.
  Interventions: Drug: Defactinib; Drug: Cetuximab; Drug: Avutometinib
- Expansion (Experimental): If you are enrolled in the Expansion, you will receive avutometinib at the recommended dose that was found in Safety Run In.
  Interventions: Drug: Defactinib; Drug: Cetuximab; Drug: Avutometinib

INTERVENTIONS:
Drug: Defactinib — Given by PO
Drug: Cetuximab — Given by IV
  Other Names: ERBITUX
Drug: Avutometinib — Given by PO

SUMMARY:
To learn if avutometinib in combination with defactinib and cetuximab can help to control unresectable, anti-EGFR-refractory, advanced colorectal cancer.

DETAILED DESCRIPTION:
The primary objective is to assess the antitumor activity of the treatment combinations based on Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1.

Secondary Objectives:

1. Assess impact of treatment combinations on survival
2. Characterize the safety profile of the treatment combinations (DLTs)
3. Evaluate the pharmacodynamics of the avutometinib combination with defactinib plus cetuximab.
4. Evaluate for pERK and Ki67 inhibition

Exploratory Objectives

* Assess blood- and tissue-based predictive biomarkers of activity upon treatment with cetuximab plus avutometinib plus defactinib
* Demonstrate feasibility of establishing patient-derived xenograft (PDX) models in matched patients with cetuximab-refractory mCRC to evaluate for biomarkers of response and mechanisms of resistance.
* Explore mechanisms of resistance to cetuximab plus avutometinib and defactinib

ELIGIBILITY:
Inclusion Criteria:

• Provision of signed Informed Consent prior to any screening procedures being performed.

* Non-English speaking participants will be eligible for participation with involvement of the MD Anderson Language Assistance department in the informed consent process (per MD Anderson SOP 04_Informed Consent Process).
* Individuals lacking the ability, based on reasonable medical judgment, to understand and appreciate the nature and consequences of participation in this study will not be eligible for participation.

  * Age ≥ 18 years at the time of informed consent.
  * Histologically (or cytologically) confirmed diagnosis of adenocarcinoma of the colon or rectum, with clinical confirmation of unresectable and/or metastatic disease that is measurable according to RECIST1.1 criteria.
  * Mutation status at the time of colorectal cancer diagnosis performed on tumor tissue or circulating tumor

DNA (prior to any anti-EGFR directed therapy):

* KRAS, NRAS, EGFR ectodomain, BRAF V600E wild-type status

  * Prior treatment with at least one systemic chemotherapy regimen for mCRC, or recurrence/progression with development of unresectable or metastatic disease within 6 months of adjuvant chemotherapy for resected colorectal cancer.
  * Prior treatment with:
* anti-EGFR therapy (cetuximab or panitumumab) setting for at least 16 weeks with either CR or PR as best response, prior to progression • ECOG performance status ≤ 1.

  • Participants who received chemotherapy must have recovered (Common Terminology Criteria for Adverse Events [CTCAE] Grade ≤1) from the acute effects of chemotherapy except for residual alopecia or Grade 2 peripheral neuropathy prior to day 1 of study. A washout period of at least 21 days is required between last chemotherapy dose and day 1 of study (provided the patient did not receive radiotherapy).

  • Participants who received radiotherapy must have completed and fully recovered from the acute effects of radiotherapy. A washout period of at least 7 days is required between end of radiotherapy and day 1 of study.

  • Adequate hematologic status: Absolute neutrophil count (ANC) ≥ 1.5 x 109/L; Hemoglobin (Hgb) ≥ 9 g/dL with or without transfusions; Platelets (PLT) ≥ 100 x 109/L without transfusions

  • Adequate liver function:
* ALT and AST ≤3 × ULN, or ≤5 × ULN in the presence of liver metastases
* Total bilirubin ≤ 1.5 × ULN and < 1.5 mg/dL
* Note: Participants with hyperbilirubinemia due to non-hepatic cause (e.g., hemolysis, hematoma) may be enrolled following discussion and agreement with the principal investigator. • Adequate renal function: Serum Creatinine ≤ 1.5 x ULN, or calculated creatinine clearance (measured via 24-hour urine collection) ≥ 40 mL/min at screening

  * QTc interval ≤ 480 ms (preferably the mean from triplicate ECGs)
  * Able to take oral medications.
  * Because the teratogenicity of cetuximab is not known, the participant, if sexually active, must be postmenopausal, surgically sterile, or using effective contraception (hormonal or barrier methods). Female participants of childbearing potential must have a negative serum pregnancy test within 7 days prior to enrollment
  * Willing and able to participate in the trial and comply with all trial requirements.
  * Participants with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational agent may be included after consultation with the medical monitor.

Exclusion Criteria:

1. History of grade 3 or 4 allergic reaction or intolerability attributed to cetuximab or panitumumab.
2. History of allergic reactions attributed to compounds of chemical or biologic composition similar to those of cetuximab, or if the patient had red meat allergy/tick bite history.
3. Previously exposed to ERK1/2, MEK or BRAF inhibitor
4. Any known symptomatic brain metastasis
5. Note: Participants previously treated or untreated for this condition who are asymptomatic in the absence of corticosteroid and anti-epileptic therapy are allowed. Known brain metastases must be stable for ≥ 4 weeks, with imaging (e.g., magnetic resonance imaging [MRI] or computed tomography [CT]) demonstrating no current evidence of progressive brain metastases at screening.
6. Known leptomeningeal disease
7. A history or current evidence/risk of retinal vein occlusion (RVO) or central serous retinopathy (CSR).
8. Previous or concurrent malignancy within 3 years of study entry, with the following exceptions: adequately treated basal or squamous cell skin cancer, superficial bladder cancer, prostate intraepithelial neoplasm, carcinoma in-situ of the cervix, or other noninvasive or indolent malignancy; other solid tumors treated curatively without evidence of recurrence for at least 3 years prior to study entry.
9. Impaired cardiovascular function or clinically significant cardiovascular diseases, including any of the following:

1. History of acute coronary syndromes (including myocardial infarction, unstable angina, coronary artery bypass grafting, coronary angioplasty, or stenting) <12 months prior to screening, 2. Symptomatic chronic heart failure (i.e., Grade 2 or higher), history or current evidence of clinically significant cardiac arrhythmia and/or conduction abnormality <6 months prior to screening except atrial fibrillation and paroxysmal supraventricular tachycardia, 3. The participant has a personal history of any of the following conditions: syncope of cardiovascular etiology, ventricular arrhythmia of pathological origin (including, but not limited to, ventricular tachycardia and ventricular fibrillation), or sudden cardiac arrest.

4. Uncontrolled hypertension defined as persistent elevation of systolic blood pressure ≥ 170 mmHg or diastolic blood pressure ≥ 100 mm Hg, despite current therapy.

10. The participant has active systemic bacterial or fungal infection (requiring intravenous (IV) antibiotics and/or antifungals at time of initiating study treatment).

11. Know Human Immunodeficiency Virus (HIV) that is active and or/requires therapy 12. Active hepatitis B or hepatitis C infection

1. Active HBV is defined as any of the following: i) HBsAg(+), HBV DNA >200 IU/mL (36 copies/mL) ii) HBsAg(+), HBV DNA ≤200 IU/mL and persistent or intermittent elevation of ALT/AST and/or liver biopsy showing chronic hepatitis with moderate or severe necroinflammation. iii) Note: Participants who are HBsAg(-), HBcAb(+) are eligible and should be monitored/treated as per local standard of care. 2. Active HCV is defined as: i) HCV antibody positive; AND ii) Presence of HCV RNA. 13. Impaired gastrointestinal function or disease that may significantly alter the absorption of study drug (e.g., ulcerative diseases, uncontrolled vomiting, malabsorption syndrome, small bowel resection with decreased intestinal absorption).

14. Any other condition that would, in the Investigator's judgment, contraindicate the participant's participation in the clinical study due to safety concerns or compliance with clinical study procedures.

15. Major surgery ≤ 6 weeks prior to starting study drug or failure to recover from side effects of such procedure at the discretion of the treating investigator.

16. Systemic anti-cancer therapy within 4 weeks of the first dose of study intervention or within 5 half-lives of the previous drug, whichever is longer.

17. Pregnant or nursing (lactating) women, where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive hCG laboratory test.

18. History of Rhabdomyolysis 19. Medical, psychiatric, cognitive or other conditions that may compromise the patient's ability to understand the participant information, give informed consent, comply with the study protocol or complete the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Estimated)
Dates: Start 2025-02-24 (Actual); Primary Completion 2029-02-01 (Estimated); Study Completion 2029-02-01 (Estimated)

PRIMARY OUTCOMES:
Safety and adverse events (AEs) | Through study completion; an average of 1 year.
  Incidence of Adverse Events, Graded According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version (v) 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Christine Parseghian, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org